CLINICAL TRIAL: NCT01877876
Title: Assessing the Accuracy of the RevK Sensor for Non-Invasive Hemoglobin Monitoring
Brief Title: Assessing the Accuracy of the RevK Sensor
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 10-00524E
Record Dates: First submitted 2013-05-28; First posted 2013-06-14 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Patients Undergoing Spine Surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient undergoing spine surgery

SUMMARY:
Evaluation of a new generation of sensors for monitoring blood hemoglobin. The newest version is RevK.

DETAILED DESCRIPTION:
Evaluation of a new generation of sensors for monitoring blood hemoglobin with the Masimo non-invasive hemoglobin monitor. The newest sensor version is RevK.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female
* American Society of Anesthesiology Classification 1, 2 or 3
* Scheduled to undergo spine or hip surgery

Exclusion Criteria:

* Pregnant or nursing
* Patients who in the study investigators clinical judgement would not be suitable for research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To assess the accuracy of the RevK sensor for measuring blood hemoglobin compared to a laboratory-derived hemoglobin value. | Intermittently during spine surgery
  Primary outcome is based on the difference between a value from the SpHb (Masimo SpHb™ continuous hemoglobin reading) minus tHb (laboratory hemoglobin determination).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald D Miller, MD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States